CLINICAL TRIAL: NCT07106216
Title: Evaluating Two Novel Near-infrared Spectroscopy Devices for Non-invasive Monitoring of Traumatic Brain Injury in the Neuro Critical Care Unit.
Brief Title: Evaluating Near-infrared Spectroscopy Devices for Monitoring Traumatic Brain Injury
Acronym: NIRS in TBI
Status: Not yet recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Brain Physics Laboratory, Division of Neurosurgery, Department of Clinical Neurosciences, University of Cambridge, UK (Unknown); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Peter J. Hutchinson MD, Professor, University of Cambridge
Other Study IDs: IRAS 330193; EP/S022139/1 (Other Grant/Funding Number: EPSRC)
Record Dates: First submitted 2025-05-14; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Tramatic Brain Injury
Keywords: brain; head; injury; severe; nirs
MeSH Terms: conditions — Wounds and Injuries; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe brain injury: Those with severe (as defined by the Glasgow Coma Scale) brain injuries

SUMMARY:
This project seeks to evaluate the capabilities of new Near Infrared Spectroscopy (NIRS) devices, which use light to measure brain activity, for monitoring how the brain and body react after a serious head injury (TBI), particularly in the immediate and shortly following periods. Data recorded from these devices will help determine if they can effectively monitor additional complications and outcomes in adults over 18 with severe TBIs in a specialised intensive care unit for brain injuries (NCCU) at Addenbrooke's Hospital (Cambridge, UK). We will use two different NIRS devices similar to those currently used in the NCCU but with extra improvements. Both devices are proven to be safe and do not require surgery or internal procedures.

Participants will be recruited based on several criteria and monitored early in their NCCU admission. Monitoring will be daily for 6 hours, lasting from half a week to two weeks, depending on recovery progress. After the initial 10 patients, we will perform an interim analysis and may adjust the recording duration. We aim to recruit a maximum of 50 participants in total. Due to their condition, participants will not be able to give permission to participate, so we will seek it from their next of kin within 24 hours of admission. The study will only observe and not influence treatment. We will also collect additional clinical data, such as scans, the patient's condition six months after the injury, and other medical information for analysis.

The data collection period for this study will last up to 2 years. We will remove any personal details from the patient data. The body function data, with personal details removed, will be transferred and stored on the Brain Physics Lab server (segregated) and University of Cambridge computers for analysis. Any data not saved in dedicated long-term storage will be deleted after use.

DETAILED DESCRIPTION:
This study will apply novel near-infrared spectroscopy (NIRS) devices within the neurocritical care unit (NCCU) in Addenbrooke's Hospital (Cambridge, UK). The devices are non-invasive and are shown to be safe. The study is expected to last around year. It will not be used to inform treatment, and patient care is to remain identical regardless of study inclusion.

This study will use two NIRS devices, both of which have enhancements over systems used within the NCCU currently. We aim to develop NIRS-based biomarkers that could be used to support the treatment of those suffering from traumatic brain injury (TBI).

Upon receiving advice from the patient's consultee, the participant will be recorded with two different NIRS devices for a total of six hours daily (three hours per device). Recordings will occur daily for the duration of the participant's admission to the NCCU. We request access to clinical data, for example, blood pressure, heart rate, injuries suffered, CT and MRI scans and six-month outcomes for analytical purposes. As the devices are light-based, skin tone or ethnicity data is requested as is age-band for subject-specific modelling. This data will then be used to develop metrics based on existing literature that describe the brain health of the participant.

Participants will be unable to provide informed consent. Therefore, we will seek advice from their next of kin or in the event they cannot be identified within 24 hours, the treating clinician.

Participants will be those in the NCCU. They will be suffering from moderate or severe TBI. It is very likely they will be in an unconscious state. The study is limited to adults (defined as ≥18 years of age).

Two devices are planned for use in this study. The first device is a Lumo (Gowerlabs Ltd, UK), a high-density diffuse optical tomography device. This device is a modified version of a CE-marked device. The second is a custom broadband NIRS device that has met all legal and regulatory requirements. It is assembled out of CE-marked components although the device itself is not CE-marked.

We aim to start patient recordings to start in Q2 2025. The maximum number of participants for this study is set to 50. The end date is set at the 31st of December 2025.

By recording with these devices, we hope to develop new methods for monitoring TBI- an injury that impacts tens of millions annually. The novelty of this study comes from the devices applied. They have only been applied in a limited context previously within TBI cohorts, although are common in research. This study will be used to inform future studies which we hope will ultimately lead to improved patient care.

ELIGIBILITY:
Inclusion Criteria:

Those in the Neuro Critical Care Unit at Addenbrooke's (Cambridge, UK) AND

Patients with moderate or severe head trauma AND

Over 18 AND

Those with intracranial pressure monitoring probes."

Exclusion Criteria:

We will not monitor anyone aged under 18 OR

We will not monitor anyone with penetrating wounds in the area we want to monitor OR

Patients who are enrolled on >2 other research studies, as per local guidelines OR

Moribund at presentation OR

Those with infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Addenbookes (Cambridge, UK) neuro critical care ward patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Score Extended | 6 months after admission
  The Glasgow Outcome Scale-Extended (GOSE) is a detailed assessment tool used to evaluate the functional status and recovery of patients following traumatic brain injury (TBI), categorizing outcomes into eight levels ranging from death to full recovery. It helps clinicians and researchers understand the long-term impact of TBI on a patient's daily life and guides treatment and rehabilitation efforts. Lower numbers are worse (1=dead). Higher numbers are better (8=Good recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Smielewski, PhD, Study Director — Cambridge University Hospitals

IPD SHARING:
Plan to Share IPD: No
We do not have permission to share IPD

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT07106216/SAP_000.pdf